CLINICAL TRIAL: NCT04660903
Title: Treatment of Fistula in Ano With Autologous Fatty Tissue Cells Transplantation
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Severe adverse reaction on patient
Sponsor: Konstantinos Tsimogiannis (Other)
Responsible Party: Sponsor-Investigator, Konstantinos Tsimogiannis, Consultant, Uppsala University Hospital
Organization: Uppsala University Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Fettcell studie
Record Dates: First submitted 2020-11-22; First posted 2020-12-09 (Actual); Last update posted 2022-06-13 (Actual); Status verified 2022-06

CONDITIONS: Fistula in Ano; Transsphincteric Anal Fistula
MeSH Terms: conditions — Rectal Fistula

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): One arm study - the intervention arm is the only actual
  Interventions: Procedure: Autologous fat cell transplantation

INTERVENTIONS:
Procedure: Autologous fat cell transplantation — Up to 75 ml of fatty tissue mixture fluid

SUMMARY:
This is a prospective interventional study on the treatment of transsphincteric fistula in ano. After abdominal or thigh liposuction, fat was injected around the fistula tract that was then transected percutaneously with a sharp cannula and fat injected between and around the cut parts. The internal opening was closed with a suture. Minimum follow up of 12 months is planed

DETAILED DESCRIPTION:
The study is intended to be carried out at the Department of Surgery of Uppsala University Hospital, as a single-center study. All (consecutive) otherwise healthy patients between the ages of 18-70 who have been diagnosed with perianal fistula where attempts to close the fistula is considered appropriate are asked to participate. This is done by the examining physician at their visit at the outpatient clinic. These are either patients who already have a relieving seton or those who need to be revised and treated with a seton before final closure.

They receive written information about the study plan and have time to think about it. If they choose to participate in the study, they are planed for a visit to one of the surgeons involved in the study and here get another opportunity to ask questions and then also sign an informed consent. This step can be adjusted as telephone contact due to the Covid-19 pandemic. Thereafter, they are included in the study.

The participants are operated on only by the surgeons involved, all of whom have undergone practical training in how fat cell transplantation is carried out according to the standardized Coleman method.

The procedure itself then takes place as a day surgery operation at the Samariter Hemmet ( part of the Surgical Department, Uppsala University Hospital ) operating department and either as a one- or two-step procedure, depending on whether they have a relieving seton or not. The seton has to be placed sometime before the definitive fatty tissue procedure so that there is no sign of inflammation/infection.

A 3- and 12-months follow up visit is then arranged. In these visits, the patients are examined for evaluation of the result, possible residual fistulas, and complications. Wexner score and VAS scale are filed in and saved in their patient files.

ELIGIBILITY:
Inclusion Criteria:

* Verified perianal or rectovaginal fistula
* Healthy individuals that can be accepted for an elective operation with total anesthesia.
* Signed consent

Exclusion Criteria:

* Patients under the age of 18 or over the age of 75 years
* Another disease that can affect the perianal are or the procedure
* Patients that are not able to understand and sign the consent themselves.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-10-01 (Actual); Primary Completion 2023-10-30 (Estimated); Study Completion 2024-02-28 (Estimated)

PRIMARY OUTCOMES:
Clinical healing of fistula in ano | 3 months after index operation
  No fistula opening and no fistula related symptoms on clinical examination and with anal ultrasound at the outpatient clinic
Clinical healing of fistula in ano | 12 months after index operation
  No fistula opening and no fistula related symptoms on clinical examination and with anal ultrasound at the outpatient clinic
Postoperative complication | 3 months after index operation
  Possible complications linked to index operation
Postoperative complication | 12 months after index operation
  Possible complications linked to index operation

SECONDARY OUTCOMES:
Functional effects | 3 months after index operation
  Incontinence or constipation after index operation that will be assessed with Wexner score ( On a scale of 0-20, with 0 = perfect continence and 20 = complete incontinence ).
Functional effects | 3 months after index operation
  Studied with a calendar with stool frequency and consistency, filled by patients for descriptive analysis
Functional effects | 12 months after index operation
  Incontinence or constipation after index operation that will be assessed with Wexner score ( On a scale of 0-20, with 0 = perfect continence and 20 = complete incontinence )
Functional effects | 12 months after index operation
  Studied with a calendar with stool frequency and consistency, filled by patients for descriptive analysis
Injected fat quantity | During index operation
  The quantity of fat cell mixture injected per patient
Visual Analog Pain Scale score | 3 months after index operation
  Pain or discomfort after the treatment, using Visual analog scale, for the first 3 weeks of the postoperative period. The scale ranges from 0 8 no pain ) to 10 ( maximum possible pain )
Visual Analog Pain Scale score | 12 months after index operation
  Pain or discomfort after the treatment, using Visual analog scale, for the first 3 weeks of the postoperative period. The scale ranges from 0 8 no pain ) to 10 ( maximum possible pain )

CONTACTS AND LOCATIONS:
Overall Officials: Wilhelm Graf, Professor, Study Director — Uppsala University
Locations (1):
- Uppsala University Hospital, Uppsala, Sweden

IPD SHARING:
Plan to Share IPD: No
Not allowed by the ethical committee and data legislations. If this is required, completion of the Ethical decision is needed

REFERENCES:
- [Background] Choi S, Ryoo SB, Park KJ, Kim DS, Song KH, Kim KH, Chung SS, Shin EJ, Cho YB, Oh ST, Kang WK, Kim MH. Autologous adipose tissue-derived stem cells for the treatment of complex perianal fistulas not associated with Crohn's disease: a phase II clinical trial for safety and efficacy. Tech Coloproctol. 2017 May;21(5):345-353. doi: 10.1007/s10151-017-1630-z. Epub 2017 May 31. PMID 28567691
- [Background] Norderval S, Lundby L, Hougaard H, Buntzen S, Weum S, de Weerd L. Efficacy of autologous fat graft injection in the treatment of anovaginal fistulas. Tech Coloproctol. 2018 Jan;22(1):45-51. doi: 10.1007/s10151-017-1739-0. Epub 2017 Dec 28. PMID 29285682
- [Background] Herreros MD, Garcia-Arranz M, Guadalajara H, De-La-Quintana P, Garcia-Olmo D; FATT Collaborative Group. Autologous expanded adipose-derived stem cells for the treatment of complex cryptoglandular perianal fistulas: a phase III randomized clinical trial (FATT 1: fistula Advanced Therapy Trial 1) and long-term evaluation. Dis Colon Rectum. 2012 Jul;55(7):762-72. doi: 10.1097/DCR.0b013e318255364a. PMID 22706128
- [Background] Dozois EJ, Lightner AL, Mathis KL, Chua HK, Kelley SR, Fletcher JG, Dietz AB, Friton JJ, Butler GW, Faubion WA. Early Results of a Phase I Trial Using an Adipose-Derived Mesenchymal Stem Cell-Coated Fistula Plug for the Treatment of Transsphincteric Cryptoglandular Fistulas. Dis Colon Rectum. 2019 May;62(5):615-622. doi: 10.1097/DCR.0000000000001333. PMID 30664554
- [Background] Pu LLQ, Coleman SR, Cui X, Ferguson REH Jr, Vasconez HC. Autologous fat grafts harvested and refined by the Coleman technique: a comparative study. Plast Reconstr Surg. 2008 Sep;122(3):932-937. doi: 10.1097/PRS.0b013e3181811ff0. PMID 18766062
- [Background] Borowski DW, Gill TS, Agarwal AK, Tabaqchali MA, Garg DK, Bhaskar P. Adipose Tissue-Derived Regenerative Cell-Enhanced Lipofilling for Treatment of Cryptoglandular Fistulae-in-Ano: The ALFA Technique. Surg Innov. 2015 Dec;22(6):593-600. doi: 10.1177/1553350615572656. Epub 2015 Feb 20. PMID 25710946